CLINICAL TRIAL: NCT00657618
Title: Department of Defense Protocol for the Use of Sodium Stibogluconate (Pentostam) as a Treatment for Leishmaniasis
Brief Title: Use of Sodium Stibogluconate as a Treatment for Leishmaniasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-12631; WU#04-19011 (Other: IRB); Pentostam (Registry Identifier: NCT00657618)
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Leishmaniasis
Keywords: Leishmaniasis, Sodium stibogluconate, Pentostam, sand fly
MeSH Terms: conditions — Leishmaniasis | interventions — Antimony Sodium Gluconate; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment only (Experimental): All consented subjects who meet all inclusion and no exclusion criteria will enter this open label protocol and be treated with Sodium Stibogluconate (SSG).
  Interventions: Drug: Sodium Stibogluconate (SSG)

INTERVENTIONS:
Drug: Sodium Stibogluconate (SSG) — 100 mg/ml/vial. Treatment for laboratory-confirmed leishmaniasis with SSG 20mg/kg/d intravenously (IV) for 10 days or 20 days; visceral leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days as a second line of therapy for those failing or intolerant of Ambisome; and mucosal leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days.
  Other Names: Pentostam (GlaxoSmithKline)

SUMMARY:
Leishmanias is a disease caused by the bite of sandflies and is found in many parts of the world including the Europe, Southwest Asia, Africa and the Middle East. This disease is a threat for military soldiers in areas where this disease is found. Sodium stibogluconate (SSG) or Pentostam (Glaxo Smith Kline, United Kingdom) is an Investigational New Drug (IND) product used by the Department of Defense for over 20 years to treat cutaneous, mucosal and visceral leishmanias. This drug is not licensed for commercial use in the United States because of very limited need for the product in the U.S.A. The primary objective of this protocol is to collect safety data on the use of Pentostam for treatment of laboratory-confirmed leishmaniasis with SSG 20mg/kg/d IV for 10 days or 20 days and visceral and mucocutaneous leishmaniasis with SSG 20mg/kg/d IV for 28 days.

Due to low enrollment, the protocol was later amended in version 11 submitted 19May2010 in serial no. 0096) to remove the efficacy objective and only collect safety data for enrolled subjects. Prior to this amendment, data were entered on case report forms (CRFs). Per the Sponsor's discretion, CRFs were no longer required and protocol-specified treatment details and safety assessments were recorded in the patients' medical records (study file) only. No data entry or statistical analyses of patient data was conducted.

DETAILED DESCRIPTION:
Leishmaniasis is a protozoal disease transmitted by sandflies and is endemic in many parts of the world including Central and South America, Europe, Southwest Asia, Africa, and the Middle East. Infected humans may develop cutaneous (Old or New World), mucocutaneous (New World), or visceral leishmaniasis. The disease is a medical threat for military soldiers assigned in endemic areas and currently a major cause of morbidity in soldiers deployed to the Middle East and a complication of military exercises in Panama, Honduras, and South America. Sodium stibogluconate (SSG) is an Investigational New Drug (IND) product that has been in use by the Department of Defense (DoD) for over 20 years for the treatment of cutaneous, mucosal and visceral leishmaniasis. The primary objective of this protocol is to treat laboratory-confirmed leishmaniasis with SSG 20mg/kg/d intravenously (IV) for 10 days or 20 days; visceral leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days as a second line of therapy for those failing or intolerant of Ambisome; and mucosal leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days. Subjects will be monitored daily and outcome measured at the end of therapy by the degree of healing of cutaneous lesions or resolution of laboratory abnormalities and symptoms in the case of mucosal and visceral leishmaniasis.

Pentavalent antimonials (Pentostam, Glaxo Smith Kline, United Kingdom) has been used to treat leishmaniasis for more than 50 years. This drug has not been licensed for commercial use in the United States, likely because of limited commercial marketability. Worldwide and within the DoD, there is a great deal of experience and use of Pentostam for the treatment of leishmaniasis. SSG is a pentavalent antimony (Sb) complexed to a carbohydrate whose exact structure and mechanism of action are not known. It is provided as a 100 mg antimony/mL solution that contains a preservative, m-chlorocresol. The kidneys excrete most of the dose within 24 hours. In 1984, the World Health Organization recommended the daily dose of antimony in the treatment of visceral leishmaniasis to be increased to 20 mg/kg/day. A randomized controlled trial of 40 subjects with American, New World, cutaneous leishmaniasis (ACL) found 100% cure rates with 20 mg/kg/day Sb for 20 days but only a 76% cure if 10 mg/kg/day for 10 days was used. A comparison of three treatment schedules in 36 subjects with CL (single rapid infusion, continuous 24 hour infusion, or every eight hour doses) found no advantage over using once daily dosing. A review of the controlled trials of SSG concludes that a recommended course of therapy is 20 mg/kg/day with no upper limit to dose for 20 days for CL and 20 mg/kg/day for 28 days for visceral or mucocutaneous leishmaniasis. The Pentostam® package insert suggests that 10-20 mg/kg/day with a maximum dose of 850 mg for a minimum of 20 days be used; however, based on the Centers for Disease Control and Prevention (CDC) and Walter Reed Army Medical Center (WRAMC) experience and their practice guidelines, 20 mg/kg/day with no upper limit to dosage is used. In this protocol there will be no upper limit to the dose. WRAMC recently published their CL treatment experience primarily in New World leishmaniasis comparing SSG 20 mg/kg for 10 or 20 days and found 100% of volunteers in the 10-day group were cured. In this study 15% were Leishmania major infections. Comparable results are expected for Old World leishmaniasis based on clinical experience and current literature.

Detailed toxicity data for the 20 mg/kg/day dose are provided by several studies. Percentages from the WRAMC experience are included here. Subjective musculoskeletal complaints are common (58%), as well as elevated hepatocellular (67%) and pancreatic enzyme levels (97%) and nonspecific electrocardiogram (EKG) changes (T wave changes). These side effects are usually reversible, and no deaths have been associated with SSG at WRAMC. Other SSG toxic effects include headache (22%), rash (9%), thrombocytopenia, depression of various hematologic cell lines (44%), phlebitis, anaphylaxis, inflammation around lesions, and transient coughing after infusion. Other associated symptoms include anorexia, malaise, myalgia, abdominal pain, headache, lethargy, sweating, vertigo, facial flushing, initial worsening of skin lesions, epistaxis, jaundice and peripheral neuropathy. In our above-mentioned 10 versus 20 days study, the adverse events (AE) were significantly decreased in the cohort receiving the 10 days versus 20 with myalgias in 42% (versus 68%), with less chemical pancreatitis and fewer hematologic parameter disorders. Angioedema during SSG infusion has recently been described in two subjects at WRAMC. Both subjects responded quickly to benadryl treatment without complications. Both subjects were subsequently skin tested with SSG intradermally for hypersensitivity and one reacted.

Alternative heat therapies have been used to successfully treat CL. Laboratory investigation showed that Leishmania infection is sensitive to heat. Various forms of heat application in human CL has shown variable efficacy. The TTI Thermomed™ device is currently U.S. Food and Drug Administration (FDA), section 510-K cleared for use in the treatment of CL. This device uses localized current field radio frequency. Other therapies that may be effective for treating CL include topical paromomycin and oral fluconazole.

ELIGIBILITY:
Inclusion Criteria:

1. DoD healthcare beneficiary of any age and gender.
2. Clinicoepidemiologic or parasitologic diagnosis (microscopy, PCR or culture) of Leishmania infection.
3. Able to provide informed consent or assent (children).
4. All participants (both male and female) must agree to take precautions not to become pregnant or father a child for at least 2 months after receiving SSG.

Exclusion Criteria:

1. Pregnancy. Females of childbearing potential must have negative urine human chorionic gonadotropin hormone (HCG) within 96 hours start of infusion period.
2. History of hypersensitivity to pentavalent antimonials.
3. Any of the following on screening examination:

   1. QTc interval greater or equal to 0.5 sec
   2. Severe cardiac disease (disabling valvular heart disease, myopathy, or arrhythmias)
   3. History of recurrent pancreatitis
   4. Liver failure or active hepatitis with transaminases > 3x upper limit of normal
   5. Renal failure or creatinine > 2.5 mg/dL
   6. Thrombocytopenia (platelets <100,000/mm^3)
   7. White blood cell count < 2000 / mm^3
   8. Hematocrit < 30 %

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roseanne Ressner, MD, Principal Investigator — Walter Reed National Military Medical Center, Infectious Disease
Locations (1):
- Walter Reed National Military Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 total patients, 74 treated, 34 completed treatment, 43 withdrawals
Pre-assignment Details: Due to low enrollment protocol was amended to remove efficacy objective and only collect safety data. No data entry or statistical analyses of patient data was conducted.
Groups:
- Sodium Stibogluconate (SSG): All consented subjects who meet all inclusion and no exclusion criteria will enter this open label protocol and be treated with Sodium Stibogluconate (SSG).
  Sodium Stibogluconate (SSG): 100 mg/ml/vial. Treatment for laboratory-confirmed leishmaniasis with SSG 20mg/kg/d intravenously (IV) for 10 days or 20 days; visceral leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days as a second line of therapy for those failing or intolerant of Ambisome; and mucosal leishmaniasis will be treated with SSG 20mg/kg/d IV for 28 days.
Period: Overall Study
Arm/Group | Sodium Stibogluconate (SSG)
Started | 77
Completed | 34
Not Completed | 43
Not completed — Adverse Event | 32
Not completed — Withdrawal by Subject | 8
Not completed — negative for leishmaniasis | 2
Not completed — didn't start due to schedule conflicts | 1

BASELINE CHARACTERISTICS:
Population: Due to low enrollment the protocol was amended to remove efficacy objective and only collect safety data for subjects. No data entry or statistical analyses of patient data was conducted.
Arm/Group | Sodium Stibogluconate (SSG)
Number analyzed (Participants) | 77
Age, Customized [Number; unit: participants] — Due to low enrollment the protocol was amended to remove efficacy objective and only collect safety data for subjects. No data entry or statistical analyses of patient data including age data was conducted. Population: Data was not collected
Sex/Gender, Customized [Number; unit: participants] — Due to low enrollment the protocol was amended to remove efficacy objective and only collect safety data for subjects. No data entry or statistical analyses of patient data including gender data was conducted. Population: Data not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Discontinued Due to Adverse Experience, by Type of Adverse Experience
Description: The safety of Pentostam (SSG) treatment was evaluated through the daily assessment of AEs during treatment. Additionally, clinical laboratory tests including serum chemistry (glucose, electrolytes, blood urea nitrogen [BUN], creatinine, alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin, alkaline phosphatase [ALK], amylase, and lipase) and hematology (hemoglobin, hematocrit, platelets, and white blood cells with differential); vital signs measurements; electrocardiograms (ECGs); and physical examinations were performed at screening and prior to Pentostam infusion on Days (± 2) 5, 10, 15, 20, 25, and 28 (Days 25 and 28 for patients with visceral or mucocutaneous leishmaniasis only). At the completion of Pentostam treatment, patients were encouraged to arrange follow-up at 2, 6, and 12 months after treatment; however, follow-up was not required.
Time Frame: prior to infusion on days (± 2) 5, 10, 15, 20, 25, and 28
Population: 74 patients received at least one dose of IV pentostam
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Only
Number analyzed (Participants) | 74
Participants
  Myalgia/arthralgia | 12
  Elevated liver-associated enzymes | 10
  Rash | 3
  Subtle elevation of amylase and lipase | 1
  Misdiagnosis | 1
  Decreased white blood cell count | 1
  Nephrotoxicity | 1
  Chemical pancresatitis | 1
  Drug reaction | 1

2. Primary Outcome: Number of Participants Experiencing Serious or Unexpected Adverse Events, by Type of Serious or Unexpected Adverse Events
Description: as for outcome 1
Time Frame: prior to infusion on days 2) 5, 10, 15, 20, 25, and 28
Population: 74 patients received at least one dose of IV pentostam
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Only
Number analyzed (Participants) | 74
Participants
  Elevated lipase level | 4
  Chemical hepatitis | 1
  Allergic reaction with atypical presentation | 1
  Misdiagnosis | 1
  Allergic reaction | 1
  Hospitalized for unhealed cutaneous lesion | 1

ADVERSE EVENTS:
Time Frame: prior to infusion on days (± 2) 5, 10, 15, 20, 25, and 28
Description: Safety of Pentostam was evaluated through daily assessment of AEs. Clinical lab tests including serum chemistry (glucose, electrolytes, blood urea nitrogen, creatinine, alanine aminotransferase, aspartate aminotransferase], total bilirubin, alkaline phosphatase], amylase, and lipase) and hematology (hemoglobin, hematocrit, platelets, and white blood cells with differential); vital signs measurements; electrocardiograms); and physical examinations were performed at screening and prior to infusion
Arm/Group | Treatment Only
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 8/74
Other Adverse Events (participants affected / at risk) | 32/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Only (N=74)
Elevated lipase/aysmpotmatic chemical pancreatitis (Investigations) | 4 (4)
Chemical hepatitis (Investigations) | 1 (1)
Allergic reaction with atypical presentation (Immune system disorders) | 1 (1)
Misdiagnosis (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Hospitalization for unhealed lesion (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Only (N=74)
Myalgia/arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12)
Elevated liver-assocated enzymes (Investigations) | 10 (10)
Rash (Immune system disorders) | 3 (3)
Subtle ECG changes (Investigations) | 1 (1)
Elevation of amylase and lipase (Investigations) | 1 (1)
Misdiagnosis (Investigations) | 1 (1)
Decreased white blood cell count (Investigations) | 1 (1)
Nephrotoxicity (Investigations) | 1 (1)
Chemical pancreatitis (Gastrointestinal disorders) | 1 (1)
Drug reaction (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to low enrollment protocol was amended to remove efficacy objective and only collect safety data. No data entry or statistical analyses of patient data was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No